CLINICAL TRIAL: NCT00067262
Title: A Double-Blind, Placebo-Controlled Trial to Evaluate the Safety and Efficacy of Depakote ER for the Treatment of Bipolar Disorder in Children and Adolescents
Brief Title: An Outpatient Study of the Effectiveness and Safety of Depakote ER in the Treatment of Mania/Bipolar Disorder in Children and Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M01-342
Record Dates: First submitted 2003-08-13; First posted 2003-08-15 (Estimated); Last update posted 2006-08-04 (Estimated); Status verified 2006-08

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder Type 1 (manic or mixed type)
MeSH Terms: conditions — Bipolar Disorder; Mania

INTERVENTIONS:
Drug: Divalproex Sodium Extended-Release Tablets

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of Depakote ER (Divalproex Sodium Extended-Release Tablets) compared to placebo in the treatment of bipolar disorder, manic or mixed type in children and adolescents ages 10-17 years.

ELIGIBILITY:
INCLUSION CRITERIA

* Current primary diagnosis of bipolar I disorder, mania or mixed type
* Outpatient between 10 and 17 years of age
* Young Mania Rating Scale score greater than or equal to 20 during screening/washout and at Day 1

EXCLUSION CRITERIA

* Axis I other than Attention Deficit Hyperactivity Disorder (ADHD), Obsessive Compulsive Disorder (OCD), Oppositional Defiant Disorder (ODD), Conduct Disorder (CD), Panic Disorder; or Axis II (e.g., personality disorder) that would interfere with compliance or confound interpretation of study results
* Current manic episode is drug-induced or secondary to a medical disorder (e.g., anti-depressants, hyperthyroidism)
* Expected to require hospitalization for the current manic episode
* Participation in psychotherapy that was started within the past 3 months, or if any significant changes are anticipated
* Has taken atomoxetine or has taken allowed stimulant medication that has not been stable for at least 3 months prior to Day 1, or a dosage adjustment is expected during the study, or that may worsen mood symptoms
* Unable to swallow tablets
* Has received depot psychoactive medication within one inter-injection interval of Day 1
* Urine toxicology screen is positive for phencyclidine (PCP), opiates, cocaine, barbiturates, benzodiazepines or amphetamines
* History of alcohol or substance dependence within past 3 mos. or substance abuse within past month
* History of failed treatment on adequate Depakote (DR or ER) for a manic episode within past 12 months
* Has taken Depakote (DR or ER) regularly for the current manic episode
* Has serious violent, homicidal, or suicidal ideation

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150
Dates: Start 2003-03

PRIMARY OUTCOMES:
Change from baseline to the final evaluation in Y-MRS score.

SECONDARY OUTCOMES:
Vital signs
Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information, Study Director — Abbott
Locations (16):
- United States (16):
  - Stanford University, Stanford, California
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Altamonte Springs, Florida
  - Professional Clinical Research, Inc., Miami, Florida
  - Segal Institute for Clinical Research, North Miami, Florida
  - Mountain West Clinical Trials, Boise, Idaho
  - Capstone Clinical Research, Libertyville, Illinois
  - Cientifica Inc at Praire View, Inc., Newton, Kansas
  - Lexington, Kentucky
  - LSU - Health Science Center, New Orleans, Louisiana
  - Brentwood Research Institute, Shreveport, Louisiana
  - New Oakland Child/Adoles and Family Center, Clinton Township, Michigan
  - Mercy Health Research, Chesterfield, Missouri
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas Medical Branch, Houston, Texas

REFERENCES:
- [Derived] Wagner KD, Redden L, Kowatch RA, Wilens TE, Segal S, Chang K, Wozniak P, Vigna NV, Abi-Saab W, Saltarelli M. A double-blind, randomized, placebo-controlled trial of divalproex extended-release in the treatment of bipolar disorder in children and adolescents. J Am Acad Child Adolesc Psychiatry. 2009 May;48(5):519-532. doi: 10.1097/CHI.0b013e31819c55ec. PMID 19325497